CLINICAL TRIAL: NCT03791242
Title: A Prospective, Randomized, Multi-center Comparative Effectiveness Study of Apnea-Hypopnea Index Using CPAP or CPAP Plus Ketogenic Diet for Treatment of Obstructive Sleep Apnea in Patients Scheduled for Bariatric Surgery
Brief Title: Ketogenic Diet and CPAP Previous Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gianfranco Silecchia, MD PhD Prof. G. Silecchia, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0199138/2018
Record Dates: First submitted 2018-12-28; First posted 2019-01-02 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Obstructed Sleep Apnea Syndrome in Patient Candidate to Baratric Surgery
MeSH Terms: interventions — Continuous Positive Airway Pressure; Diet, Ketogenic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): 33 morbidly obese patients with severe OSAS and suitable for gastric bypass surgery, who underwent 4 weeks of CPAC treatment (these patients will not be required to change their eating habits) according to the standard
  Interventions: Device: Cpap and ketogenic diet
- Group 2 (Active Comparator): 33 morbidly obese patients with severe OSAS and BS candidates who underwent CPAC + KMED treatment for 4 weeks
  Interventions: Device: Cpap and ketogenic diet

INTERVENTIONS:
Device: Cpap and ketogenic diet — Patients with severe OSAS who are BS candidates will be treated with CPAP only at night (Group 1), or CPAP at night + KMED daily (Group 2), for 4 weeks

SUMMARY:
Obstructive Sleep Apnea Syndrome (OSAS) and obesity tend to coexist and are often associated with arterial hypertension, dyslipidaemia, and insulin resistance [1]. Polysomnography (PSG) is the standard technique for diagnosing OSAS and determining its severity [2]. The results of the examination provide the Apnea-Hypopnea Index [AHI], or the Respiratory Disturbance Index [RDI]), which will be used to quantify apnea and classify its severity based on an international score. In general, an AHI scoring less than 5 is considered "normal" (5-15 mild sleep apnea; >15 moderate sleep apnea; ≥30 severe sleep apnea).

In order to improve those parameters in obese patients who have been diagnosed with OSAS and are candidates for BS (BS), national and international guidelines recommend preoperative CPAP (Continuous Positive Airway Pressure) treatment in order to reduce anaesthesia risks [3-6]. Furthermore, several studies report that obese OSAS patients benefit from preoperative weight loss [1,7] (in terms of AHI index, night snoring and arterial hypertension).

Obese patients who are candidates for BS often go on a preoperative diet in order to decrease weight and liver volume (especially of the left lobe) and correct any vitamin/mineral deficiency. The results of a recently published study show that 4 weeks of Ketogenic Micronutrient Enriched Diet (KMED) significantly reduce body weight, liver lobe volume and vitamin/mineral deficiencies in obese patients who prepare to undergo BS [8], with resulting foreseeable reduction of intraoperative complications and surgical time.

To date, there are no prospective multicenter randomized trials demonstrating whether a preoperative ketogenic diet associated with CPAP use improves OSAS versus treatment with CPAP alone, with the possibility of reducing the preoperative treatment period.

Aim of the study: To assess the clinical advantage in combining two preoperative strategies (CPAP + KMED) compared to preoperative treatment with CPAP alone, for the reduction of surgical risks in morbidly obese patients with severe OSAS who are scheduled for BS.

DETAILED DESCRIPTION:
A recent clinical study published in 2014 on the New England Journal of Medicine found that often even an initial modest body weight reduction can favourably modify apnea events and severity during the night, with the latter that can be reduced by about 30% (AHI) for a 10% weight reduction compared to the initial weight [1]. However, considering the average AHI data reported by the authors, which do not include post-treatment information, statistical elements at our disposal are insufficient to assess the "effect size". Therefore, a sample of 65 patients per group will be needed for the evaluation of the primary endpoint (statistical significance of 5% [two-tailed], 80% power, "effect size" 0.25, calculated using the G* Power software, Düsseldorf, Germany). A total of 66 patients will be enrolled (22 patients per participating site) on the baseline assumption of a dropout of 10%. Most drop-outs may result from CPAP use and, in particular, discomfort experienced by the patient with tube and facial mask, difficult acceptance because of psychological reasons (shame or negative expectations in terms of partner judgment), or subjective feeling of claustrophobic suffocation or anxiety. The expected drop-out for KMED with the Ketocompleat protocol is 15%. Indeed, in Schiavo et al [8] study, most patients (86%) showed high acceptability of the Ketocompleat ketogenic protocol prescribed in the four weeks of preoperative treatment, and the only side effect reported was mild headache with associated modest halitosis, especially during the initial treatment days, which, however, did not prevent patients from continuing with the protocol.

Experiment design and patient randomization

Spontaneous, prospective, comparative and multicentre trial including 66 patients with severe OSAS (polysomnogram with AHI≥30) suitable for gastric bypass surgery, and randomized into 2 groups:

GROUP 1: 33 morbidly obese patients with severe OSAS and suitable for gastric bypass surgery, who underwent 4 weeks of CPAC treatment (these patients will not be required to change their eating habits) according to the standard; GROUP 2: 33 morbidly obese patients with severe OSAS and BS candidates who underwent CPAC + KMED treatment for 4 weeks.

Randomization will be conducted via permuted-block design (PBD), with stratification of patients based on age, gender, and enrollement site Preoperative ketogenic micronutrient-enriched diet: The ketogenic diet has been used for many years in clinical settings [9]. Given its safety and effectiveness in determining weight loss, associated with optimal adherence and patient compliance, the ketogenic diet has recently been used by several obesity surgery centers in the preoperative management of obese patients who are candidates for BS [8, 10-11]. The validated Ketocompleat protocol [8] will serve as the KMED of choice. In particular, the protocol will provide a diet with ketogenic characteristics that patients will have to follow for breakfast, snack, lunch and snack, and replacement of the evening meal with the Ketocompleat ketogenic supplement. Figure 1 shows a daily diet sample.

In short, to ensure that all patients follow the same diet, the investigator will use the software (https://www.eatthismuch.com) to develop two ketogenic diet plans (plan 1, days 1-14; plan 2, days 15-28), containing specific amounts of foods to be consumed. Each ketogenic plan will comprise: 1150 to 1250 kcal/day, of which 4% carbohydrates, 71% fat, and 25% proteins. The composition of the supplement to use for the trial (Ketocompleat, MVMedical Solutions, Serravalle, Republic of San Marino) is shown in Table 1. Ketocompleat is a supplement included in the Ministry of Health's food supplement register (code 94721); given its carbohydrate-free formulation, it can easily be associated to a low-carbohydrate ketogenic diet. The diet plans and the Ketocompleat supplement will be provided free of charge to all trial participants by MVMedical Solutions, which will have no role in designing trial and patient enrollement in the different participating sites, or in processing any trial-related data.

Patient adherence to the prescribed preoperative diet will be confirmed through the following scientifically validated tests: 3-Day Estimated Food and Records and 72-h Recalls [8], while the presence of ketone bodies in the urine (Ketur-Test, Roche Diagnostic, Milan, Italy) associated with weight loss will be used as the patient compliance index. The Ketur test will be performed in outpatient mode during the weekly diet check.

Polysomnography

Polysomnography is a sleep study that collects a variety of parameters and conditions, such as oxygen saturation, heart rate, presence (or absence in the case of apnea) of airflow through mouth and nose, presence (or absence) of thoracic and abdominal movements, position held by the subject during sleep, and snoring during sleep. By analysing these data, it will be possible to define: number of episodes of haemoglobin desaturation during sleep (desaturation index per hour - ODIindex), presence or absence of apnea during sleep, differentiating between true apnea true (absence of air flow) and hypopneas (air flow present, though substantially reduced), determination of "obstructive" "central" or "mixed" apnea/hypopnea, hourly frequency of apnea/ hypopnea ( apnea/hypopnea events per hour or AHI index), which allows defining the degree of severity of the disorder (disease stage), AHI in supine and non-supine position (often this datum documents greater apnea frequency in the supine position compared to data relating to the patient in lateral decubitus), and snoring time during sleep. In order to evaluate the clinical advantage offered by the combination of the two preoperative strategies (CPAP and ketogenic diet therapy) compared to CPAP preoperative treatment alone, for the reduction of the surgical risk in morbidly obese OSAS BS candidates, patients of both groups will undergo polysomnography before the trial and after 4 weeks of CPAP alone or combined CPAP + KMED treatment. The tolerance interval for PSG execution at the end of the treatment is 7 days; otherwise, patients will be considered drop-outs.

CPAP-type ventilator prescription CPAP use is the gold standard for the treatment of sleep apnea syndrome. The CPAP device consists of a small fan connected to the patient through a tube and a facial mask (nasal or oronasal). This device provides continuous air flow that maintains the airways open, preventing the collapse (closing) of the critical points responsible for respiratory obstruction during sleep, thus avoiding or limiting sleep apnea. Patients with severe OSAS who are BS candidates will be treated with CPAP only at night (Group 1), or CPAP at night + KMED daily (Group 2), for 4 weeks.

Preoperative investigations and after 4 weeks of CPAP or CPAP + KMED treatment

In the BS Centers participating in the trial, both experimental groups will undergo the following evaluation:

* Complete blood count with WBC differential, triglycerides, total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, GOT, GPT, ΥGT, nitrogen, creatinine, urea, iron, ferritin, ketone bodies, baseline glucose, baseline insulin, and CRP
* Body weight, height and BMI calculation
* Waist and hip circumference
* Chest X-ray
* Blood gas analysis
* Spirometry
* Polysomnography

Laboratory/instrumental clinical analyses, polysomnography and CPAP will be performed in the sites participating in the project; data obtained will be evaluated by a Pneumologist, while the statistical analysis will be entrusted to a Biostatistician.

Inclusion criteria: patients of both sexes with BMI ≥35 with severe OSAS; age between 18-65 years; non-smokers or who have quit smoking for at least 3 months.

Exclusion criteria: kidney and/or liver conditions that would make a KMED diet unsuitable (creatinine levels >1.8 mg/dL or liver enzyme levels (glutamic pyruvic transaminase [GPT] or glutamic oxaloacetic transaminase [GOT]) less than three times over the upper normal threshold, and psychological problems that would make CPAP treatment problematic. Patients with obesity >60 BMI.

Primary endpoint: evaluate the effect of combined (CPAP + KMED) therapy vs CPAP on the AHI after 4 weeks. Secondary end points: evaluate CRP levels, arterial pressure and lipid panel (total cholesterol, HDL, LDL and triglycerides) in the two study groups.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥35 Kg/m2
* Severe OSAS
* Non-smokers or who have quit smoking for at least 3 months

Exclusion Criteria:

* kidney and/or liver conditions that would make a KMED diet unsuitable (creatinine levels >1.8 mg/dL or liver enzyme levels (glutamic pyruvic transaminase [GPT] or glutamic oxaloacetic transaminase [GOT]) less than three times over the upper normal threshold
* psychological problems that would make CPAP treatment problematic
* BMI > 60 Kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index | 0 - 4 weeks
  evaluate the effect of combined (CPAP + KMED) therapy vs CPAP on the AHI after 4 weeks

SECONDARY OUTCOMES:
Blood exam | 0 - 4 weeks
  C-reactive protein

OTHER OUTCOMES:
Arterial Pressure | 0 - 4 weeks
  arterial pressure measure
Blood exam | 0 - 4 weeks
  Lipid pattern

CONTACTS AND LOCATIONS:
Locations (1):
- ICOT Hospital, Latina, Italy

IPD SHARING:
Plan to Share IPD: Undecided